CLINICAL TRIAL: NCT01376362
Title: The Treatment of Macular Edema Secondary to Uveitis Using Topical Interferon Gamma
Brief Title: Topical Interferon Gamma for Macular Edema Secondary to Uveitis
Acronym: JakStat2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Nida Sen, Principal Investigator, NEI, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110167; 11-EI-0167 (Other: CNS IRB)
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-09

CONDITIONS: Anterior Uveitis; Uveitis
Keywords: Cystoid Macular Edema; Intermediate Uveitis; Uveitis; OCT; Interferon-Gamma (IFN-Gamma)
MeSH Terms: conditions — Uveitis, Anterior; Uveitis; Macular Edema; Uveitis, Intermediate | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interferon gamma-1b (Experimental): Interferon gamma-1b (Actimmune®, InterMune, Inc, Brisbane, CA 94005) was supplied to participants in single-use dropperettes. Each dropperette contained approximately 0.2 mL of interferon gamma-1b (Actimmune®). Participants received 28 dropperettes at the baseline visit and were instructed to place four drops (approximately 7 μg per drop) topically on the cornea of the study eye four times per day for seven days.
  Interventions: Drug: Interferon Gamma-1b

INTERVENTIONS:
Drug: Interferon Gamma-1b — Interferon gamma-1b (Actimmune®, InterMune, Inc, Brisbane, CA 94005) was supplied to participants in single-use dropperettes. Each dropperette contained approximately 0.2 mL of interferon gamma-1b (Actimmune®). Participants received 28 dropperettes at the baseline visit and were instructed to place four drops (approximately 7 μg per drop) topically on the cornea of the study eye four times per day for seven days.
  Other Names: Actimmune®

SUMMARY:
The objective of this study is to investigate the safety and efficacy of ocular instillations of interferon gamma-1b as a potential treatment for cystoid macular edema (CME) secondary to uveitis.

DETAILED DESCRIPTION:
Objective: Information gathered from NEI laboratories suggests that cystoid macular edema (CME) is caused by the disequilibrium of the JakStat and mTor signal transduction pathways in the retinal pigment epithelium (RPE). We wish to investigate whether stimulating the JakStat pathway with topically applied interferon gamma-1b can be a therapeutic intervention for the treatment of CME secondary to uveitis. The objective of this study is to investigate the safety and efficacy of ocular instillations of interferon gamma-1b as a potential treatment for CME secondary to uveitis.

Study Population: Five participants with CME as evidenced by OCT (> 275 microns central macular thickness and/or loss of foveal contour) secondary to uveitis will receive topical ocular instillations of interferon gamma-1b. Up to seven participants may be enrolled in order to obtain the five participants to be included in the analysis if participants withdraw prior to receiving interferon gamma-1b.

Design: This Phase I/II, non-randomized, prospective, uncontrolled, single-center study will involve instilling four drops of interferon gamma-1b (approximately 30 μg) topically on the cornea of the study eye four times a day for one week and measuring the potential response with optical coherence tomography (OCT).

Outcome Measures: The primary outcome is the change in excess central macular thickening as measured by OCT in response to interferon gamma-1b. Treatment success is defined as a 25% decrease in excess central macular thickening at Week 1 as compared with baseline. Secondary efficacy outcomes include changes in macular volume as measured by OCT, visual acuity, intraocular pressure and intraocular inflammation as graded upon slit lamp examination. Secondary safety outcomes include ocular surface irritation assessed by fluorescein staining of the cornea and conjunctiva to assess toxicity, the number and severity of systemic and ocular toxicities, the number of adverse events and the proportion of participants with a visual loss of ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters.

ELIGIBILITY:
Inclusion Criteria

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol's informed consent document.
3. Participant has a diagnosis of CME (central thickness of >275 microns on OCT and/or disruption of foveal contour) secondary to uveitis in at least one eye (the study eye).
4. Participant is willing to comply with the study procedures and is expected to be able to return for all study visits.
5. Participant has visual acuity of 20/400 or better in the study eye.
6. Female participants of childbearing potential must not be pregnant or breast-feeding.
7. Both female participants of childbearing potential and male participants able to father a child must agree to practice two acceptable forms of contraception during the study and for six weeks following the last administration of investigational product. Acceptable methods of contraception include hormonal contraception (i.e., birth control pills, injected hormones dermal patch or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation or vasectomy).

Exclusion Criteria

1. Participant is unable to tolerate the ocular instillations or follow study procedures.
2. Participant has a significant active infection (an infection requiring treatment as determined by the medical team) that in the principal investigator's best medical judgment would preclude participation.
3. Participant has multiple sclerosis (MS), as interferon gamma may cause MS exacerbations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Nida Sen, MD, MHSc, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Battle TE, Lynch RA, Frank DA. Signal transducer and activator of transcription 1 activation in endothelial cells is a negative regulator of angiogenesis. Cancer Res. 2006 Apr 1;66(7):3649-57. doi: 10.1158/0008-5472.CAN-05-3612. PMID 16585190
- [Background] Khorana HG. Rhodopsin, photoreceptor of the rod cell. An emerging pattern for structure and function. J Biol Chem. 1992 Jan 5;267(1):1-4. No abstract available. PMID 1730574
- [Background] Shi G, Maminishkis A, Banzon T, Jalickee S, Li R, Hammer J, Miller SS. Control of chemokine gradients by the retinal pigment epithelium. Invest Ophthalmol Vis Sci. 2008 Oct;49(10):4620-30. doi: 10.1167/iovs.08-1816. Epub 2008 Apr 30. PMID 18450597

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interferon Gamma-1b
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age Continuous [Median (Full Range); unit: years] | 55 (12.51) [32 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Excess Central Macular Thickening in the Study Eye, as Measured by Optical Coherence Tomography (OCT), at Week One Compared to Baseline
Description: Central macular thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
µm | -38.60 (130.26) [-102 to 54]

2. Secondary Outcome: Change in Excess Central Macular Thickening in the Fellow Eye, as Measured by Optical Coherence Tomography (OCT), at Week One Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
µm | 12.00 (29.12) [0 to 36]

3. Secondary Outcome: Change in Excess Central Macular Thickening in the Study Eye, as Measured by Optical Coherence Tomography (OCT), at Week Two Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline and 2 Weeks
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
µm | -47.40 (85.96) [-106 to 108]

4. Secondary Outcome: Change in Excess Central Macular Thickening in the Fellow Eye, as Measured by Optical Coherence Tomography (OCT), at Week Two Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline and 2 Weeks
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
µm | 30.20 (64.43) [-16 to 84]

5. Secondary Outcome: Change in Macular Volume in the Study Eye, as Measured by Optical Coherence Tomography (OCT), at Week One Compared to Baseline
Description: Macular volume was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
mm^3 | -0.02 (0.36) [-0.60 to 0.40]

6. Secondary Outcome: Change in Macular Volume in the Fellow Eye, as Measured by Optical Coherence Tomography (OCT), at Week One Compared to Baseline
Description: as for outcome 5
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
mm^3 | 0.14 (0.21) [-0.10 to 0.40]

7. Secondary Outcome: Change in Macular Volume in the Study Eye, as Measured by Optical Coherence Tomography (OCT), at Week Two Compared to Baseline
Description: as for outcome 5
Time Frame: Baseline and 2 Weeks
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
mm^3 | 0.00 (0.32) [-0.30 to 0.50]

8. Secondary Outcome: Change in Macular Volume in the Fellow Eye, as Measured by Optical Coherence Tomography (OCT), at Week Two Compared to Baseline
Description: as for outcome 5
Time Frame: Baseline and 2 Weeks
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
mm^3 | 0.06 (0.34) [-0.30 to 0.40]

9. Secondary Outcome: Change in ETDRS Best-corrected Visual Acuity (BCVA) in the Study Eye at Week One Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
ETDRS Letters | 0.20 (5.63) [-7 to 6]

10. Secondary Outcome: Change in ETDRS Best-corrected Visual Acuity (BCVA) in the Fellow Eye at Week One Compared to Baseline
Description: as for outcome 9
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
ETDRS Letters | 1.60 (4.72) [-1 to 10]

11. Secondary Outcome: Change in ETDRS Best-corrected Visual Acuity (BCVA) in the Study Eye at Week Two Compared to Baseline
Description: as for outcome 9
Time Frame: Baseline and 2 Weeks
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
ETDRS Letters | 4.00 (9.03) [-10 to 13]

12. Secondary Outcome: Change in ETDRS Best-corrected Visual Acuity (BCVA) in the Fellow Eye at Week Two Compared to Baseline
Description: as for outcome 9
Time Frame: Baseline and 2 Weeks
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
ETDRS Letters | 3.20 (6.87) [-2 to 15]

13. Secondary Outcome: Change in Intraocular Pressure (IOP) in the Study Eye at Week One Compared to Baseline
Description: Intraocular pressure was recorded using a standard Goldmann applanation tonometer, a device for the measurement of intraocular pressure between 0 to 78 mm Hg.
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
mm Hg | 0.40 (2.07) [-2 to 3]

14. Secondary Outcome: Change in Intraocular Pressure (IOP) in the Fellow Eye at Week One Compared to Baseline
Description: as for outcome 13
Time Frame: Baseline and 1 Week
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
mm Hg | -1.60 (7.02) [-14 to 3]

15. Secondary Outcome: Change in Intraocular Pressure (IOP) in the Study Eye at Week Two Compared to Baseline
Description: as for outcome 13
Time Frame: Baseline and 2 Weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
mm Hg | 0.40 (1.34) [-1 to 2]

16. Secondary Outcome: Change in Intraocular Pressure (IOP) in the Fellow Eye at Week Two Compared to Baseline
Description: as for outcome 13
Time Frame: Baseline and 2 Weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
mm Hg | -2.20 (7.40) [-15 to 4]

17. Secondary Outcome: Proportion of Participants With a Visual Loss of 15 or More Early Treatment Diabetic Retinopathy Study (ETDRS) Letters in the Study Eye
Description: as for outcome 9
Time Frame: Baseline and 2 Weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
Percentage of Participants | 0

ADVERSE EVENTS:
Arm/Group | Interferon Gamma-1b
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No